CLINICAL TRIAL: NCT04111718
Title: The Impact of Procedural Awareness of Knee Injections for Osteoarthritis on Patient Perceptions of Effectiveness
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: ArthroBiologix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ABx-prp-001
Record Dates: First submitted 2019-09-30; First posted 2019-10-01 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Viewing of preparation (Experimental): The patient will be in the room for the preparation of the PRP and will receive a description of the centrifuge process from the physician administering the injection.
  Interventions: Biological: Platelet-rich plasma (PRP); Behavioral: Viewing of preparation
- Blinded to preparation (Sham Comparator): The patient will leave the room after their blood is drawn and will not view the preparation of the PRP, and will also not receive a description of the centrifuge process.
  Interventions: Biological: Platelet-rich plasma (PRP)

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP) — Autologous platelet-rich plasma which will be derived from blood drawn from the patient.
Behavioral: Viewing of preparation — The patient will receive a description of the preparation process and will view the preparation in the centrifuge.
  Arms: Viewing of preparation

SUMMARY:
The purpose of this study is to determine whether outcomes for patients receiving intra-articular platelet-rich plasma (PRP) injections for knee osteoarthritis are influenced by observation of the preparatory steps to the procedure. The viewing of the steps involved in the administration of PRP may increase the effectiveness of the treatment in comparison to patients who have not observed the preparatory steps.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women ages 50-80 years
* Diagnosis of symptomatic osteoarthritis of the knee based on clinical and radiographic criteria
* Provision of informed consent

Exclusion Criteria:

* Patients with inflammatory osteoarthritis
* Open wounds or sores over the knee joint
* Patients that will likely have problems, in the judgement of the investigators, with maintaining follow-up

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
VAS Pain | 12 weeks
  Visual analog scale pain on a 0-10 scale, with higher scores indicating worse pain.

SECONDARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | 12 weeks
  Patient reported knee osteoarthritis index with subscores of pain, function and stiffness. The range of scores on the WOMAC is from 0-96, with higher scores indicating worse outcomes. The subscore of pain is on a scale of 0-20, the subscore of stiffness is 0-8, and the subscale of function is 0-68. The scores of the subscales are summed in order to get the total score.
Range of motion | 12 weeks
  Range of motion in the knee from full extension to full flexion.
Short Form 12 (SF-12) Functional outcome assessment | 12 weeks
  Health-related quality of life measure on a scale from 0-100, where higher scores indicate better function.

CONTACTS AND LOCATIONS:
Overall Officials: Moin Khan, FRCSC, Principal Investigator — McMaster University
Locations (1):
- ArthroBiologix, Hamilton, Ontario, Canada